CLINICAL TRIAL: NCT01135511
Title: A Phase II, Prospective, Randomized, Double Masked/Investigator Masked, Vehicle And Comparator (Sodium Hyaluronate Eye Drops) Controlled, Dose Ranging Study Of CP-690,550 Eye Drops In Subjects With Dry Eye Disease
Brief Title: A Phase II, Dose Ranging Study Of CP-690,550 Eye Drops In Patients With Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3921072
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-03

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment 1 (Experimental)
  Interventions: Drug: CP-690,550 Eye drops
- Treatment 2 (Experimental)
  Interventions: Drug: CP-690,550 Eye drops
- Treatment 3 (Experimental)
  Interventions: Drug: CP-690,550 Eye drops
- Treatment 4 (Placebo Comparator)
  Interventions: Drug: CP-690,550 Eye drops-vehicle
- Treatment 5 (Active Comparator)
  Interventions: Drug: Sodium Hyaluronate

INTERVENTIONS:
Drug: CP-690,550 Eye drops — Ophthalmic topical solution, low dose, dosed once/day, 8 weeks
  Arms: Treatment 1
Drug: CP-690,550 Eye drops — Ophthalmic topical solution, medium dose, dosed once/day, 8 weeks
  Arms: Treatment 2
Drug: CP-690,550 Eye drops — Ophthalmic topical solution, high dose, dosed once/day, 8 weeks
  Arms: Treatment 3
Drug: CP-690,550 Eye drops-vehicle — Ophthalmic topical solution, vehicle, dosed once/day, 8 weeks
  Arms: Treatment 4
Drug: Sodium Hyaluronate — Ophthalmic topical solution, dosed 6 times/day, 8 weeks
  Arms: Treatment 5

SUMMARY:
The purpose of the study is to evaluate dose-response, efficacy and safety of CP-690,550 eye drops in patients with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjective symptoms of dry eye for at least 6 months
* Signs of moderate to severe dry eye (corneal staining score and schirmer test without anesthesia)

Exclusion Criteria:

* Women who are nursing, pregnant or planning pregnancy during the study
* Participation in other studies within 30 days of screening visit
* Ocular disorders that may confound interpretation of study results

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- Japan (22):
  - Pfizer Investigational Site, Ichinomiya, Aichi-ken
  - Pfizer Investigational Site, Narashino, Chiba
  - Pfizer Investigational Site, Urayasu, Chiba
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Chiba, Japan
  - Pfizer Investigational Site, Tokyo, Japan
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Yokohama, Kangawa
  - Pfizer Investigational Site, Kyoto, Kyoto
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Fuji, Shizuoka
  - Pfizer Investigational Site, Numazu, Shizuoka
  - Pfizer Investigational Site, Shizuoka, Shizuoka
  - Pfizer Investigational Site, Susono, Shizuoka
  - Pfizer Investigational Site, Chiyoda-ku, Tokyo
  - Pfizer Investigational Site, Hamura, Tokyo
  - Pfizer Investigational Site, Minato-ku, Tokyo
  - Pfizer Investigational Site, Ohta-ku, Tokyo
  - Pfizer Investigational Site, Sumida-ku, Tokyo
  - Pfizer Investigational Site, Tachikawa, Tokyo
  - Pfizer Investigational Site, Taito-ku, Tokyo
  - Pfizer Investigational Site, Tokyo
- South Korea (2):
  - Pfizer Investigational Site, Gwangju
  - Pfizer Investigational Site, Seoul

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921072&StudyName=A%20Phase%20II%2C%20Dose%20Ranging%20Study%20Of%20CP-690%2C550%20Eye%20Drops%20In%20Patients%20With%20Dry%20Eye%20Disease

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, during the 2-week run-in period, enrolled participants were administered artificial tears 4 times daily after signing informed consent.
Groups:
- CP-690,550 Eye Drops Vehicle Group in Japan; CP-690,550 Eye Drops Vehicle Group in Korea: At baseline (Day 0), the participants were administered the first dose of CP-690,550 eye drops vehicle. Participants instilled CP-690,550 eye drops vehicle with 1 drop per time and once daily during the 8-week treatment period. Participants continued to use artificial tears 4 times daily during the treatment period.
- CP-690,550 Eye Drops 0.001% Group in Japan; CP-690,550 Eye Drops 0.001% Group in Korea: At baseline (Day 0), the participants were administered the first dose of CP-690,550 eye drops 0.001%. Participants instilled CP-690,550 eye drops 0.001% with 1 drop per time and once daily during the 8-week treatment period. Participants continued to use artificial tears 4 times daily during the treatment period.
- CP-690,550 Eye Drops 0.003% Group in Japan; CP-690,550 Eye Drops 0.003% Group in Korea: At baseline (Day 0), the participants were administered the first dose of CP-690,550 eye drops 0.003%. Participants instilled CP-690,550 eye drops 0.003% with 1 drop per time and once daily during the 8-week treatment period. Participants continued to use artificial tears 4 times daily during the treatment period.
- CP-690,550 Eye Drops 0.005% Group in Japan; CP-690,550 Eye Drops 0.005% Group in Korea: At baseline (Day 0), the participants were administered the first dose of CP-690,550 eye drops 0.005%. Participants instilled CP-690,550 eye drops 0.005% with 1 drop per time and once daily during the 8-week treatment period. Participants continued to use artificial tears 4 times daily during the treatment period.
- Sodium Hyaluronate Eye Drops 0.1% Group in Japan: At baseline (Day 0), the participants were administered the first dose of sodium hyaluronate eye drops 0.1% and could instill sodium hyaluronate eye drops 0.1% up to 6 times a day (including the first dose). Participants instilled sodium hyaluronate eye drops 0.1% with 1 drop per time and 6 times daily for 8 weeks.
Period: Overall Study
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan | CP-690,550 Eye Drops Vehicle Group in Korea | CP-690,550 Eye Drops 0.001% Group in Korea | CP-690,550 Eye Drops 0.003% Group in Korea | CP-690,550 Eye Drops 0.005% Group in Korea
Started | 41 | 42 | 41 | 40 | 39 | 21 | 19 | 21 | 21
Completed | 41 | 39 | 33 | 37 | 38 | 20 | 18 | 20 | 20
Not Completed | 0 | 3 | 8 | 3 | 1 | 1 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — could not visit the clinic | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — noncompliance with study drug taken | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan | CP-690,550 Eye Drops Vehicle Group in Korea | CP-690,550 Eye Drops 0.001% Group in Korea | CP-690,550 Eye Drops 0.003% Group in Korea | CP-690,550 Eye Drops 0.005% Group in Korea | Total
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39 | 21 | 19 | 21 | 21 | 285
Age, Customized [Number; unit: participants]
  Between 18 and 44 years | 14 | 14 | 11 | 11 | 11 | 5 | 8 | 7 | 3 | 84
  Between 45 and 64 years | 9 | 14 | 12 | 16 | 14 | 10 | 8 | 13 | 10 | 106
  >=65 years | 18 | 14 | 18 | 13 | 14 | 6 | 3 | 1 | 8 | 95
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 39 | 37 | 33 | 34 | 20 | 16 | 20 | 19 | 250
  Male | 9 | 3 | 4 | 7 | 5 | 1 | 3 | 1 | 2 | 35

OUTCOME MEASURES:

1. Primary Outcome: Changes in Corneal Staining Scores for Study Eye From Baseline at Week 8
Description: Based on the National Eye Institute (NEI) dry eye clinical trials workshop, the cornea was divided into 5 different zones. Each corneal zone was graded independently using a 0 to 3 grading scale:0=none, 1=slight, 2=moderate, 3=severe. Sum of scores of each zone led to total score. Total score range: 0 to 15, higher score indicated greater staining. Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
  Change: score at observation minus score at baseline. Negative change from baseline indicated improvement.
Time Frame: Baseline, Week 8
Population: Intent-to-treat population: Participants who received at least 1 dose of study treatment. A last observation carried forward (LOCF) was used to impute missing data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan | CP-690,550 Eye Drops Vehicle Group in Korea | CP-690,550 Eye Drops 0.001% Group in Korea | CP-690,550 Eye Drops 0.003% Group in Korea | CP-690,550 Eye Drops 0.005% Group in Korea
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39 | 21 | 19 | 21 | 21
Units on a scale | -3.0 (2.1) | -3.0 (2.8) | -3.0 (2.5) | -3.1 (2.6) | -3.2 (2.4) | -2.4 (2.4) | -3.0 (2.7) | -2.8 (1.9) | -2.2 (2.5)

2. Secondary Outcome: Changes in Corneal Staining Scores for Study Eye From Baseline
Description: as for outcome 1
Time Frame: Baseline, Week 1, 2 and 4
Population: Intent-to-treat population: Participants who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Units on a scale
  Week 1 | -2.1 (1.9) | -1.9 (2.1) | -1.9 (2.1) | -1.6 (2.0) | -2.0 (2.0)
  Week 2 | -2.4 (1.8) | -2.4 (2.0) | -3.2 (1.8) | -3.0 (2.0) | -2.8 (2.1)
  Week 4 | -2.7 (2.0) | -3.0 (2.7) | -3.2 (2.4) | -3.3 (2.5) | -2.6 (2.1)

3. Secondary Outcome: Percentage of Participants Demonstrating 100 Percent Clearing of Corneal Staining for Study Eye
Description: Percentage of participants demonstrating corneal staining score = 0 which indicates no damage in corneal surface.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
Time Frame: Week 1, 2, 4 and 8
Population: Intent-to-treat population: Participants who received at least 1 dose of study treatment. A last observation carried forward (LOCF) was used to impute missing data at Week 8.
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Percentage of participants
  Week 1 (n=41, 41, 40, 40, 39) | 4.9 | 2.4 | 5.0 | 0 | 0
  Week 2 (n=40, 41, 39, 40, 39) | 2.5 | 2.4 | 5.1 | 7.5 | 2.6
  Week 4 (n=41, 40, 35, 40, 38) | 12.2 | 5.0 | 8.6 | 7.5 | 2.6
  Week 8 (n=41, 41, 40, 40, 39, LOCF) | 12.2 | 4.9 | 7.5 | 7.5 | 0

4. Secondary Outcome: Changes in Conjunctival Staining Scores (Interpalpebral) for Study Eye From Baseline
Description: Based on the Oxford grading system, the bulbar conjunctiva of each eye was divided into 2 different zones (nasal and temporal). The nasal and temporal bulbar conjunctival zones were each graded independently using a 6-point scale (0 [Absent] to 5 [Severe]). Total score ranged from 0 (Absent) to 10 (severe), higher score=higher damage to eyes due to dryness. Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
  Change = scores at observation minus score at baseline. Negative change from baseline indicated improvement.
Time Frame: Baseline, Week 1, 2, 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Units on a scale
  Week 1 (n=41, 41, 40, 40, 39) | -0.8 (1.9) | -0.7 (1.8) | -0.6 (1.3) | -1.1 (1.7) | -0.6 (1.7)
  Week 2 (n=40, 41, 39, 40, 39) | -1.0 (2.2) | -0.8 (2.0) | -0.7 (1.5) | -1.7 (2.5) | -1.0 (2.1)
  Week 4 (n=41, 40, 35, 40, 38) | -1.2 (2.2) | -1.0 (1.7) | -0.8 (1.5) | -2.0 (2.4) | -1.1 (2.2)
  Week 8 (n=41, 41, 40, 40, 39, LOCF) | -1.0 (2.3) | -1.1 (2.1) | -0.9 (1.4) | -2.0 (2.1) | -0.9 (1.8)

5. Secondary Outcome: Changes in Tear Break Up Time (TBUT) for Study Eye From Baseline
Description: TBUT is the interval between the last complete blink and the first appearance of a dry spot, or disruption in the tear film. Using a stopwatch, the time between last complete blink and first appearance of dry spot was recorded.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
  Change: value at observation minus value at baseline. Positive change from baseline indicated improvement.
Time Frame: Baseline, Week 1, 2, 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Seconds
  Week 1 (n=41, 41, 40, 40, 39) | 0.04 (0.83) | 0.43 (3.61) | 0.19 (0.76) | 0.22 (1.95) | 0.43 (3.22)
  Week 2 (n=40, 41, 39, 40, 39) | 0.09 (0.95) | -0.31 (2.84) | 0.26 (0.84) | 0.04 (1.54) | 1.72 (8.53)
  Week 4 (n=41, 40, 35, 40, 38) | -0.01 (0.92) | 0.20 (3.61) | 0.31 (0.62) | 0.46 (1.87) | 0.53 (1.42)
  Week 8 (n=41, 41, 40, 40, 39, LOCF) | -0.06 (1.13) | -0.25 (2.17) | 0.27 (0.77) | 1.00 (3.56) | 0.76 (1.38)

6. Secondary Outcome: Changes in Schirmer Test Values Without Anesthesia for Study Eye From Baseline
Description: The Schirmer test without anesthesia was used to estimate tear flow stimulated reflexly by insertion of a filter paper strip into the conjunctival sac. The length of wetting (distance from the notch) was recorded in millimeters (to the nearest 0.5 mm). If the wetting line was oblique, the halfway point was used.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
  Change: value at observation minus value at baseline. Positive change from baseline indicated improvement.
Time Frame: Baseline, Week 1, 2, 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Millimeters
  Week 1 (n=41, 41, 40, 40, 39) | 0.78 (6.07) | 0.34 (3.10) | 0.01 (2.16) | 0.08 (3.01) | 0.71 (3.99)
  Week 2 (n=40, 41, 39, 40, 39) | 0.28 (2.77) | 0.51 (3.49) | 0.28 (2.26) | 0.93 (3.56) | 1.04 (4.53)
  Week 4 (n=41, 40, 35, 40, 38) | 0.30 (3.39) | 0.49 (2.54) | 0.13 (2.28) | 1.13 (4.23) | 0.64 (3.38)
  Week 8 (n=41, 41, 40, 40, 39, LOCF) | 0.91 (5.43) | 0.10 (2.57) | 0.74 (2.46) | 0.26 (2.93) | 1.53 (5.32)

7. Secondary Outcome: Percentage of Participants Who Achieve ≥10 mm Schirmer Test Value Without Anesthesia for Study Eye
Description: The Schirmer test without anesthesia was used to estimate tear flow stimulated reflexly by insertion of a filter paper strip into the conjunctival sac. The length of wetting (distance from the notch) was recorded in millimeters (to the nearest 0.5 mm). If the wetting line was oblique, the halfway point was used.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
Time Frame: Week 1, 2, 4 and 8
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Percentage of participants
  Week 1 (n=41, 41, 40, 40, 39) | 7.3 | 4.9 | 0 | 2.5 | 7.7
  Week 2 (n=40, 41, 39, 40, 39) | 2.5 | 4.9 | 2.6 | 7.5 | 10.3
  Week 4 (n=41, 40, 35, 40, 38) | 7.3 | 5.0 | 2.9 | 7.5 | 5.3
  Week 8 (n=41, 41, 40, 40, 39, LOCF) | 9.8 | 4.9 | 2.5 | 5.0 | 12.8

8. Secondary Outcome: Number of Participants Who Increase of ≥10 mm From Baseline in Schirmer Test Value Without Anesthesia for Study Eye
Description: as for outcome 7
Time Frame: Week 1, 2, 4 and 8
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Participants
  Week 1 (n=41, 41, 40, 40, 39) | 2 | 1 | 0 | 1 | 1
  Week 2 (n=40, 41, 39, 40, 39) | 0 | 1 | 0 | 2 | 2
  Week 4 (n=41, 40, 35, 40, 38) | 1 | 0 | 0 | 2 | 1
  Week 8 (n=41, 41, 40, 40, 39, LOCF) | 3 | 0 | 0 | 1 | 3

9. Secondary Outcome: Changes in the Ocular Comfort Index (OCI) Total Score From Baseline
Description: The OCI is a validated instrument developed to measure the frequency and intensity of 6 common dry eye symptoms: dryness, grittiness, stinging, eye tiredness, pain, and itching. It contains 12 questions, each measured on a 7-point rating scale (0 [Never] to 6 [Always], or 0 [Never had it] to 6 [Severe]). Total score ranged from 0 (none) to 72 (severe symptoms). A higher score indicates more severe dry eye symptoms.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
  Change: score at observation minus score at baseline. Negative change from baseline indicated improvement.
Time Frame: Baseline, Week 1, 2, 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Units on a scale
  Week 1 (n=41, 41, 40, 40, 39) | -1.94 (5.20) | -2.00 (6.22) | -2.13 (7.92) | -4.17 (6.86) | -3.14 (7.88)
  Week 2 (n=40, 41, 40, 40, 39) | -4.16 (9.00) | -4.76 (7.63) | -3.80 (8.77) | -5.88 (6.98) | -3.40 (6.12)
  Week 4 (n=41, 40, 35, 40, 38) | -3.27 (6.95) | -4.20 (7.08) | -5.77 (9.71) | -5.74 (7.26) | -3.58 (9.85)
  Week 8 (n=41, 41, 40, 40, 39, LOCF) | -5.09 (7.74) | -4.98 (7.67) | -3.90 (9.30) | -6.87 (8.59) | -4.22 (9.53)

10. Secondary Outcome: Number of Participants Demonstrating at Least ≥3 Unit Decrease in Ocular Comfort Index (OCI) Total Score From Baseline
Description: The OCI is a validated instrument developed to measure the frequency and intensity of 6 common dry eye symptoms: dryness, grittiness, stinging, eye tiredness, pain, and itching. It contains 12 questions, each measured on a 7-point rating scale (0 [Never] to 6 [Always], or 0 [Never had it] to 6 [Severe]). Total score ranged from 0 (none) to 72 (severe symptoms). A higher score indicates more severe dry eye symptoms.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
  Change = scores at observation minus score at baseline. Negative change from baseline indicated improvement.
Time Frame: Week 1, 2, 4 and 8
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Participants
  Week 1 (n=41, 41, 40, 40, 39) | 17 | 15 | 13 | 21 | 16
  Week 2 (n=40, 41, 40, 40, 39) | 19 | 21 | 19 | 28 | 20
  Week 4 (n=41, 40, 35, 40, 38) | 23 | 23 | 21 | 26 | 16
  Week 8 (n=41, 41, 40, 40, 39, LOCF) | 25 | 26 | 22 | 26 | 16

11. Secondary Outcome: Changes in the Ocular Surface Disease Index (OSDI) Total Score From Baseline
Description: The OSDI is a validated instrument for ocular surface diseases, measuring the ocular symptoms, vision-related function, and environmental triggers.
  The 12 items of the OSDI questionnaire were graded on a scale of 0 [none of the time] to 4 [all of the time]. The total OSDI score was then calculated on the basis of the following formula: OSDI=[(sum of scores for all questions answered) × 100]/[(total number of questions answered) × 4].
  The OSDI is scored on a scale of 0 to 100, with higher scores representing greater disability.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
  Change: score at observation minus score at baseline. Negative change from baseline indicated improvement.
Time Frame: Baseline, Week 1, 2, 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Units on a scale
  Week 1 (n=41, 41, 40, 40, 39) | -0.43 (12.33) | -3.87 (12.42) | -0.67 (12.68) | -5.00 (9.13) | -2.99 (10.27)
  Week 2 (n=40, 41, 40, 40, 39) | -4.09 (13.73) | -7.04 (12.98) | -3.13 (14.45) | -6.77 (11.28) | -2.89 (11.34)
  Week 4 (n=41, 40, 35, 40, 38) | -3.18 (13.77) | -5.99 (15.78) | -4.48 (13.92) | -5.11 (14.03) | -2.56 (12.69)
  Week 8 (n=41, 41, 40, 40, 39, LOCF) | -3.88 (14.92) | -7.07 (17.88) | -0.37 (16.77) | -5.89 (14.98) | -2.68 (15.10)

12. Secondary Outcome: Changes in the Ocular Surface Disease Index (OSDI) Subscale Score From Baseline: Ocular Symptoms
Description: The OSDI is a validated instrument for ocular surface diseases, measuring the ocular symptoms, vision-related function, and environmental triggers.
  The 12 items of the OSDI questionnaire were graded on a scale of 0 [the none of time] to 4 [all of the time]. The subscale OSDI score was then calculated on the basis of the following formula: OSDI=[(sum of scores for questions 1 to 3 answered) × 100]/[(total number of questions 1 to 3 answered) × 4].
  The OSDI is scored on a scale of 0 to 100, with higher scores representing greater disability.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
  Change: score at observation minus score at baseline. Negative change from baseline indicated improvement.
Time Frame: Baseline, Week 1, 2, 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Units on a scale
  Week 1 (n=41, 41, 40, 40, 39) | -0.81 (15.90) | -4.07 (13.83) | -3.96 (13.74) | -5.00 (12.77) | -2.56 (14.70)
  Week 2 (n=40, 41, 40, 40, 39) | -4.17 (19.61) | -8.74 (18.06) | -3.75 (14.24) | -7.92 (16.01) | -3.63 (13.49)
  Week 4 (n=41, 40, 35, 40, 38) | -3.05 (18.89) | -7.50 (19.59) | -6.19 (14.05) | -5.42 (17.56) | -1.97 (15.43)
  Week 8 (n=41, 41, 40, 40, 39, LOCF) | -3.86 (19.01) | -7.72 (21.20) | -2.29 (17.29) | -6.04 (18.87) | -0.21 (15.59)

13. Secondary Outcome: Changes in the Ocular Surface Disease Index (OSDI) Subscale Score From Baseline: Vision-Related Function
Description: The OSDI is a validated instrument for ocular surface diseases, measuring the ocular symptoms, vision-related function, and environmental triggers.
  The 12 items of the OSDI questionnaire were graded on a scale of 0 [none of the time] to 4 [all of the time]. The subscale OSDI score was then calculated on the basis of the following formula: OSDI=[(sum of scores for questions 4 to 9 answered) × 100]/[(total number of questions 4 to 9 answered) × 4].
  Thus, the OSDI is scored on a scale of 0 to 100, with higher scores representing greater disability.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
  Change: score at observation minus score at baseline. Negative change from baseline indicated improvement.
Time Frame: Baseline, Week 1, 2, 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Units on a scale
  Week 1 (n=41, 41, 40, 40, 39) | -0.36 (18.75) | -4.71 (14.31) | 0.40 (17.35) | -6.55 (12.20) | -3.33 (13.41)
  Week 2 (n=40, 41, 40, 40, 39) | -2.61 (16.88) | -5.83 (15.52) | -2.29 (20.91) | -7.06 (11.87) | -2.57 (14.48)
  Week 4 (n=41, 40, 35, 40, 38) | -1.70 (16.73) | -6.52 (15.25) | -4.74 (17.82) | -4.29 (14.04) | -2.69 (15.35)
  Week 8 (n=41, 41, 40, 40, 39, LOCF) | -2.56 (19.45) | -8.29 (16.61) | -2.07 (18.71) | -4.75 (12.49) | -3.81 (17.46)

14. Secondary Outcome: Changes in the Ocular Surface Disease Index (OSDI) Subscale Score From Baseline: Environmental Triggers
Description: The OSDI is a validated instrument for ocular surface diseases, measuring the ocular symptoms, vision-related function, and environmental triggers.
  The 12 items of the OSDI questionnaire were graded on a scale of 0 [none of the time] to 4 [all of the time]. The subscale OSDI score was then calculated on the basis of the following formula: OSDI=[(sum of scores for questions 10 to 12 answered) × 100]/[(total number of questions 10 to 12 answered) × 4].
  The OSDI is scored on a scale of 0 to 100, with higher scores representing greater disability.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
  Change: score at observation minus score at baseline. Negative change from baseline indicated improvement.
Time Frame: Baseline, Week 1, 2, 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Units on a scale
  Week 1 (n=38, 37, 40, 39, 35) | 1.21 (22.11) | -4.28 (23.66) | 0.31 (22.20) | -3.53 (15.52) | -4.88 (20.32)
  Week 2 (n=37, 37, 39, 37, 37) | -6.53 (20.43) | -7.21 (25.43) | -6.20 (22.25) | -8.56 (18.66) | -4.28 (21.48)
  Week 4 (n=38, 37, 35, 37, 36) | -6.14 (23.72) | -3.15 (30.23) | -2.14 (24.88) | -9.57 (22.78) | -4.17 (23.44)
  Week 8 (n=38, 37, 40, 39, 38, LOCF) | -7.13 (22.92) | -4.05 (34.11) | 3.02 (31.76) | -8.44 (27.83) | -4.82 (24.46)

15. Secondary Outcome: Percentage of Participants Demonstrating ≥10 Unit Decrease in Ocular Surface Disease Index (OSDI) Total Score From Baseline
Description: The OSDI is a validated instrument for ocular surface diseases, measuring the ocular symptoms, vision-related function, and environmental triggers.
  The 12 items of the OSDI questionnaire were graded on a scale of 0 [none of the time] to 4 [all of the time]. The total OSDI score was then calculated on the basis of the following formula: OSDI=[(sum of scores for all questions answered) × 100]/[(total number of questions answered) × 4].
  The OSDI is scored on a scale of 0 to 100, with higher scores representing greater disability.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
Time Frame: Week 1, 2, 4 and 8
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Percentage of participants
  Week 1 (n=41, 41, 40, 40, 39) | 14.6 | 24.4 | 12.5 | 22.5 | 20.5
  Week 2 (n=40, 41, 40, 40, 39) | 32.5 | 34.1 | 27.5 | 25.0 | 20.5
  Week 4 (n=41, 40, 35, 40, 38) | 34.1 | 37.5 | 25.7 | 35.0 | 18.4
  Week 8 (n=41, 41, 40, 40, 39, LOCF) | 34.1 | 41.5 | 22.5 | 35.0 | 20.5

16. Secondary Outcome: Number of Participants Evaluable for Time to Achievement of 100% Clearing of Corneal Staining for Study Eye
Description: Based on the National Eye Institute (NEI) dry eye clinical trials workshop, the cornea was divided into 5 different zones. Each corneal zone was graded independently using a 0 to 3 grading scale. The maximum possible staining score is 15, higher score indicated greater staining.
  100% Clearing of Corneal Staining means corneal staining score = 0. Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
Time Frame: Week 8
Population: Intent-to-treat population: Participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Participants | 8 | 4 | 6 | 5 | 1

17. Secondary Outcome: Number of Participants Evaluable for Time to Achievement of ≥10 mm Schirmer Wetting Score Without Anesthesia for Study Eye
Description: The Schirmer test without anesthesia was used to estimate tear flow stimulated reflexly by insertion of a filter paper strip into the conjunctival sac.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
Time Frame: Week 8
Population: Intent-to-treat population: Participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Participants | 8 | 6 | 2 | 4 | 7

18. Secondary Outcome: Number of Participants Evaluable for Time to Achievement of ≥3 Unit Decrease in OCI Scores
Description: The OCI is a validated instrument developed to measure the frequency and intensity of 6 common dry eye symptoms: dryness, grittiness, stinging, eye tiredness, pain, and itching. It contains 12 questions, each measured on a 7-point rating scale (0 [Never] to 6 [Always], or 0 [Never had it] to 6 [Severe]). Negative change from baseline indicated improvement. Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
Time Frame: Week 8
Population: Intent-to-treat population: Participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39
Participants | 31 | 29 | 30 | 35 | 28

19. Secondary Outcome: Number of Participants With Ocular Adverse Events (AEs)by Severity
Description: Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Ocular AEs are the events which are localized in the ocular region. Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: 8 weeks
Population: Safety analysis set: Participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan | CP-690,550 Eye Drops Vehicle Group in Korea | CP-690,550 Eye Drops 0.001% Group in Korea | CP-690,550 Eye Drops 0.003% Group in Korea | CP-690,550 Eye Drops 0.005% Group in Korea
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39 | 21 | 19 | 21 | 21
Participants
  Mild | 4 | 0 | 4 | 2 | 2 | 3 | 7 | 0 | 6
  Moderate | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 6 | 4
  Severe | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0

20. Secondary Outcome: Number of Participants With Nonocular Adverse Events (AEs) by Severity
Description: Counts of participants who had treatment-emergent nonocular AEs, defined as newly occurring or worsening after first dose. Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: 8 weeks
Population: Safety analysis set: Participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan | CP-690,550 Eye Drops Vehicle Group in Korea | CP-690,550 Eye Drops 0.001% Group in Korea | CP-690,550 Eye Drops 0.003% Group in Korea | CP-690,550 Eye Drops 0.005% Group in Korea
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39 | 21 | 19 | 21 | 21
Participants
  Mild | 7 | 12 | 10 | 10 | 8 | 2 | 1 | 5 | 4
  Moderate | 1 | 0 | 2 | 0 | 0 | 3 | 1 | 4 | 2
  Severe | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Summary of Maximum Severity of Ocular Tolerability Assessments Post Baseline for Study Eye: Number of Participants in Each Severity Scale
Description: Ocular tolerability was assessed for the 5 symptoms (burning sensation, blurred vision, ocular discomfort, pain, tearing), based on a 4-point severity scale (none, minor, moderate, and severe).
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
Time Frame: 8 weeks
Population: Safety analysis set: Participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan | CP-690,550 Eye Drops Vehicle Group in Korea | CP-690,550 Eye Drops 0.001% Group in Korea | CP-690,550 Eye Drops 0.003% Group in Korea | CP-690,550 Eye Drops 0.005% Group in Korea
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 39 | 21 | 19 | 21 | 21
Participants
  None for blurring of vision | 32 | 33 | 32 | 32 | 36 | 11 | 11 | 15 | 13
  Minor for blurring of vision | 9 | 8 | 7 | 8 | 3 | 9 | 6 | 5 | 7
  Moderate for blurring of vision | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 1
  Severe for blurring of vision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  None for burning sensation | 26 | 22 | 26 | 27 | 34 | 7 | 7 | 11 | 9
  Minor for burning sensation | 15 | 19 | 14 | 12 | 4 | 10 | 10 | 9 | 10
  Moderate for burning sensation | 0 | 0 | 1 | 1 | 0 | 3 | 2 | 1 | 2
  Severe for burning sensation | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  None for ocular discomfort | 30 | 29 | 30 | 31 | 29 | 6 | 4 | 7 | 6
  Minor for ocular discomfort | 10 | 12 | 9 | 8 | 8 | 8 | 11 | 6 | 8
  Moderate for ocular discomfort | 1 | 1 | 2 | 1 | 1 | 6 | 3 | 7 | 6
  Severe for ocular discomfort | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
  None for pain | 28 | 30 | 34 | 32 | 34 | 12 | 9 | 12 | 9
  Minor for pain | 13 | 11 | 6 | 7 | 3 | 4 | 10 | 7 | 9
  Moderate for pain | 0 | 0 | 1 | 1 | 2 | 4 | 0 | 2 | 3
  Severe for pain | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  None for tearing | 40 | 38 | 39 | 37 | 36 | 15 | 15 | 18 | 19
  Minor for tearing | 1 | 3 | 2 | 3 | 3 | 6 | 4 | 3 | 2
  Moderate for tearing | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe for tearing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Other Pre Specified Outcome: Change in Expression of Inflammatory Markers on Conjunctival Cells From Baseline: Human Leukocyte Antigen-DR Antibody Bound Per Cell for Study Eye
Description: The average level of HLA-DR expression per cell was reported as HLA-DR antibody bound per cell (ABC).
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
  Change = value at observation minus value at baseline.
Time Frame: Baseline, Week 4 and 8
Population: A subset of intent-to-treat population collected impression cytology samples from both eyes at screening, week 4 and week 8.
Measure: Mean (Standard Deviation); unit: Antibodies bound per cell
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 8 | 5 | 10 | 12 | 13
Antibodies bound per cell
  Week 4 (n=7, 4, 9, 12, 8) | 1570.4 (8698.5) | -13899.5 (13383.8) | 5394.3 (10641.9) | 1573.8 (10087.5) | -1908.6 (11259.4)
  Week 8 (n=6, 4, 6, 11, 10) | -1496.5 (10426.5) | -8326.3 (11164.6) | 56.0 (5308.4) | 3431.9 (16532.5) | 1148.5 (12129.6)

23. Other Pre Specified Outcome: Change in Expression of Inflammatory Markers on Conjunctival Cells From Baseline: Percentage of Human Leukocyte Antigen (HLA)-DR Positive for Study Eye
Description: Percentage of conjunctival epithelial cells that were positive with HLA-DR expression was calculated as HLA-DR Positive.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage of positive cells
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 8 | 5 | 10 | 12 | 13
Percentage of positive cells
  Week 4 (n=7, 4, 9, 12, 8) | -10.27 (20.73) | -0.87 (18.24) | 11.51 (18.74) | -6.83 (28.64) | 18.30 (30.40)
  Week 8 (n=6, 4, 6, 11, 10) | -6.77 (18.19) | 6.65 (25.65) | 5.17 (24.73) | -1.05 (35.75) | 11.74 (24.84)

24. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Apolipoprotein C-3
Description: Analysis of biomarkers which were immune and inflammatory mediators such as cytokines, chemokines and matrix metalloproteinases.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
  Change= value at visit minus value at baseline.
Time Frame: Baseline, Week 4 and 8
Population: A subset of intent-to-treat population collected tear samples from both eyes at baseline, week 4 and week 8.
  n=number of analyzed with sufficient quantity for testing.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
ng/mL
  Week 4 (n=4, 5, 2, 4, 3) | -30.675 (78.363) | -38.540 (93.153) | -153.500 (164.756) | -6384.063 (12606.637) | 58.500 (59.729)
  Week 8 (n=4, 6, 2, 5, 3) | -39.250 (786.061) | -5.167 (33.983) | -70.800 (16.688) | -5102.010 (11352.752) | -1.300 (1.752)

25. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Interleukin-18
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=4, 5, 2, 4, 3) | 247.5 (374.7) | -73.0 (57.6) | 146.0 (206.5) | -154.6 (287.3) | 22.5 (57.1)
  Week 8 (n=4, 6, 2, 5, 3) | -81.3 (110.7) | -6.0 (186.1) | 100.0 (43.8) | 18.0 (210.9) | 51.2 (27.0)

26. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Interleukin-6
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=4, 5, 2, 4, 3) | 76.00 (140.92) | -36.80 (48.75) | 22.50 (21.92) | -19.70 (126.34) | 16.33 (34.70)
  Week 8 (n=4, 6, 2, 5, 3) | -11.00 (23.35) | 4.00 (25.49) | 139.00 (192.33) | 25.80 (141.39) | 12.00 (14.00)

27. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Interleukin-7
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=4, 5, 2, 4, 3) | 35.8 (51.6) | -6.8 (38.8) | 28.0 (22.6) | 3.5 (73.6) | 10.0 (50.7)
  Week 8 (n=4, 6, 2, 5, 3) | 14.3 (16.7) | 19.5 (30.9) | -15.0 (8.5) | -16.4 (28.6) | 25.0 (16.5)

28. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Interleukin-8
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=4, 5, 2, 4, 3) | 365.0 (348.2) | -18.8 (739.1) | -7.0 (470.9) | -1057.3 (1954.2) | 564.3 (1171.8)
  Week 8 (n=4, 6, 2, 5, 3) | -2486.3 (4656.3) | -367.8 (961.9) | -112.5 (484.4) | -471.6 (2378.4) | 305.7 (361.9)

29. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Monocyte Chemotactic Protein 1
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=4, 5, 2, 4, 3) | -168.5 (265.3) | -438.8 (962.4) | 24.5 (79.9) | -468.0 (390.6) | 26.7 (63.1)
  Week 8 (n=4, 6, 2, 5, 3) | -179.3 (144.1) | -289.7 (1205.3) | -169.5 (217.1) | 28.2 (431.0) | -14.3 (33.9)

30. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Interleukin-12 P40/P35 Heterodimer (IL-12P70)
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=4, 5, 2, 4, 3) | -5.0 (16.1) | -5.4 (17.0) | 27.0 (14.1) | -17.0 (24.9) | 3.7 (22.7)
  Week 8 (n=4, 6, 2, 5, 3) | 17.5 (21.7) | 15.8 (57.9) | 0.0 (0.0) | 1.6 (38.4) | 31.7 (23.6)

31. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Interleukin-1 Beta
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=4, 5, 2, 4, 3) | -0.05 (1.60) | -1.42 (5.22) | 2.75 (0.35) | -4.93 (10.29) | 6.03 (8.54)
  Week 8 (n=4, 6, 2, 5, 3) | -0.70 (4.97) | -0.42 (5.84) | 6.00 (8.49) | -2.14 (7.88) | 2.03 (0.15)

32. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Interleukin-1 Receptor Antagonist
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=3, 5, 2, 4, 3) | 76500.0 (363953.6) | -172800.0 (256165.4) | 269500.0 (498510.3) | -370575.0 (647507.1) | 15600.0 (156124.6)
  Week 8 (n=4, 6, 2, 5, 2) | -256000.0 (451986.0) | 153833.3 (317150.7) | 200000.0 (144249.8) | -268260.0 (546901.3) | 397550.0 (621476.1)

33. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Interleukin-23
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
ng/mL
  Week 4 (n=4, 5, 2, 4, 3) | 3.15 (6.14) | -13.80 (22.14) | 8.00 (21.21) | -7.13 (19.21) | 2.73 (3.04)
  Week 8 (n=4, 6, 2, 5, 3) | -6.78 (18.62) | 3.60 (16.65) | -4.00 (9.90) | 0.60 (6.02) | 0.00 (0.00)

34. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Matrix Metalloproteinase-3
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
ng/mL
  Week 4 (n=4, 5, 2, 4, 3) | 2.675 (5.952) | -1.948 (3.682) | -0.470 (1.598) | -24.833 (48.019) | 0.957 (1.202)
  Week 8 (n=4, 6, 2, 5, 3) | 21.205 (42.696) | -0.517 (3.527) | -0.650 (0.919) | -14.476 (31.070) | 0.203 (0.313)

35. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Matrix Metalloproteinase-9
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
ng/mL
  Week 4 (n=4, 5, 2, 4, 3) | 22.3 (35.8) | -13.2 (29.5) | 8.5 (12.0) | -88.3 (120.8) | 35.0 (60.6)
  Week 8 (n=4, 6, 2, 5, 3) | 0.0 (0.0) | 57.0 (90.1) | 37.5 (53.0) | -41.2 (46.7) | 26.7 (69.0)

36. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Vascular Endothelial Growth Factor
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=4, 5, 2, 4, 3) | 152.5 (1620.5) | -942.0 (2466.2) | 840.0 (735.4) | -1486.5 (4486.5) | 546.7 (546.4)
  Week 8 (n=4, 6, 2, 5, 3) | -1812.5 (1477.6) | 790.0 (1639.2) | -910.0 (2588.0) | 734.0 (3267.6) | -699.3 (1094.8)

37. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Alpha-1 Antitrypsin
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
ng/mL
  Week 4 (n=4, 5, 2, 4, 3) | -1115.0 (3226.2) | -4054.0 (8558.2) | 1535.0 (2170.8) | -628.5 (5314.7) | 5400.0 (3104.5)
  Week 8 (n=4, 6, 2, 5, 3) | -2902.5 (4534.4) | 505.0 (2977.2) | -1375.0 (1944.5) | 1220.8 (4111.8) | 2246.7 (2329.9)

38. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Interleukin-17A
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=4, 5, 2, 4, 3) | 1.98 (5.47) | -2.08 (4.28) | 1.95 (2.76) | -4.30 (9.40) | 1.60 (1.44)
  Week 8 (n=4, 6, 2, 5, 3) | -1.18 (1.39) | 0.88 (4.75) | 0.00 (0.00) | -3.58 (8.01) | 3.93 (4.61)

39. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Chemokine (C-X-C Motif) Ligand 10 (CXCL10) (Alias Gamma-Interferon Inducible Protein 10: IP10)
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=3, 5, 2, 4, 3) | -1196.7 (3885.1) | -7224.0 (27315.6) | 14545.0 (24967.9) | -11622.5 (28687.6) | 15103.3 (56584.3)
  Week 8 (n=4, 6, 2, 5, 2) | -13440.0 (27749.2) | 18971.7 (30883.3) | -6230.0 (7028.6) | 6306.0 (24845.5) | -9690.0 (13732.0)

40. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Chemokine (C-X-C Motif) Ligand 9 (CXCL9) (Alias Monokine Induced by Gamma Interferon: MIG)
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=3, 4, 2, 4, 3) | -633.3 (1325.5) | -47485.0 (110811.6) | 21025.0 (45078.1) | -18020.0 (44942.7) | 14003.3 (22925.3)
  Week 8 (n=4, 5, 2, 5, 2) | -34722.5 (62344.4) | 3118.0 (23681.2) | -10150.0 (2899.1) | 22148.0 (36704.1) | -4220.0 (5741.7)

41. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Chemokine ( C-C Motif) Ligand 20 (CCL20) (Alias Macrophage Inflammatory Protein 3 Alpha: MIP3A)
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=4, 5, 2, 4, 3) | 1.3 (541.7) | 47.4 (281.2) | 630.0 (325.3) | -1562.5 (2787.4) | -301.3 (1138.3)
  Week 8 (n=4, 6, 2, 5, 3) | -1237.8 (1975.3) | 534.5 (868.9) | -360.0 (1004.1) | -327.6 (2083.1) | 246.7 (331.6)

42. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Chemokine (C-C Motif) Ligand 5 (CCL5) (Alias Regulated on Activation, Normal T Cell Expressed, and Secreted: RANTES)
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=4, 5, 2, 4, 3) | 13.25 (31.28) | -12.06 (70.14) | 21.50 (40.31) | -28.98 (57.50) | 19.43 (51.60)
  Week 8 (n=4, 6, 2, 5, 3) | -61.48 (79.46) | -3.83 (81.17) | 6.50 (36.06) | -9.58 (49.45) | -8.93 (15.77)

43. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Tissue Inhibitor of Metalloproteinase 1 (TIMP-1)
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
ng/mL
  Week 4 (n=4, 5, 2, 4, 3) | 12.5 (85.9) | -19.8 (73.5) | 124.5 (173.2) | -131.8 (165.9) | 142.3 (375.9)
  Week 8 (n=4, 6, 2, 5, 3) | -48.5 (69.8) | 34.3 (75.2) | -109.0 (168.3) | -76.8 (88.1) | 114.0 (167.7)

44. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Epidermal Growth Factor
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
pg/mL
  Week 4 (n=4, 5, 2, 4, 3) | -0.5 (495.3) | -213.2 (1803.5) | -138.5 (186.0) | 0.5 (3816.2) | -121.7 (1815.2)
  Week 8 (n=4, 6, 2, 5, 3) | -15.5 (370.2) | 361.0 (857.7) | -885.0 (1322.3) | -122.0 (1612.5) | -212.7 (532.5)

45. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Albumin
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
mcg/mL
  Week 4 (n=4, 5, 2, 4, 3) | -228.00 (409.55) | -28.20 (94.15) | 42.50 (181.73) | 111.75 (293.07) | 164.67 (73.04)
  Week 8 (n=4, 6, 2, 5, 3) | 99.50 (354.15) | 125.17 (292.09) | 1.00 (147.08) | 96.00 (141.26) | 81.33 (75.63)

46. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Mucin 5AC
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Relative unit/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
Relative unit/mL
  Week 4 (n=3, 5, 2, 4, 3) | 1704.00 (4222.07) | -871.40 (4857.15) | 383.00 (24.04) | -35221.50 (67264.76) | 1651.67 (7544.36)
  Week 8 (n=4, 6, 2, 5, 3) | -18222.00 (32490.62) | 487.83 (5164.47) | 6926.00 (10004.15) | -35105.40 (84919.27) | -1698.33 (2346.05)

47. Other Pre Specified Outcome: Number of Participants Evaluated for Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Mucin 4
Description: Number of analyzed with sufficient quantity for analysis of biomarkers which were immune and inflammatory mediators such as cytokines, chemokines and matrix metalloproteinases.
  Results from study eye are reported. The study eye was defined as the eye with the worse (higher) corneal staining score at baseline.
Time Frame: Week 4 and 8
Population: A subset of intent-to-treat population collected tear samples from both eyes at baseline, week 4 and week 8.
Measure: Number; unit: Participants
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
Participants
  Week 4 | 2 | 2 | 1 | 1 | 1
  Week 8 | 0 | 2 | 1 | 1 | 1

48. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline - Mucin 16 Carbohydrate Antigen 125
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Relative unit/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
Relative unit/mL
  Week 4 (n=4, 5, 2, 4, 3) | 44.8 (337.3) | -228.6 (1493.7) | -41.0 (312.5) | -648.5 (1710.9) | 130.0 (178.0)
  Week 8 (n=4, 6, 2, 5, 3) | -487.3 (364.0) | 4.0 (910.5) | 265.5 (685.2) | -427.6 (1479.9) | -289.3 (86.8)

49. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Mucin 1
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Relative unit/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
Relative unit/mL
  Week 4 (n=4, 5, 2, 4, 3) | 41.0 (35.6) | 194.8 (428.5) | 79.5 (89.8) | -328.5 (634.9) | -5.3 (23.5)
  Week 8 (n=4, 6, 2, 5, 3) | -97.0 (183.0) | 33.5 (124.2) | 30.5 (57.3) | -80.2 (200.1) | -15.3 (23.2)

50. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Lipocalin 1
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
mcg/mL
  Week 4 (n=4, 5, 2, 4, 3) | -17.00 (2539.88) | 257.00 (382.18) | -3115.50 (4418.71) | -651.00 (659.50) | 573.00 (8434.01)
  Week 8 (n=4, 6, 2, 5, 3) | -1524.50 (2083.82) | 588.67 (1504.14) | -3560.00 (5048.74) | 222.60 (1420.46) | -417.00 (4540.91)

51. Other Pre Specified Outcome: Change in the Biomarker in Tear Fluid for Study Eye From Baseline -Total Protein
Description: as for outcome 24
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan
Number analyzed (Participants) | 17 | 14 | 9 | 8 | 11
mcg/mL
  Week 4 (n=4, 5, 2, 4, 3) | 748.8 (4116.3) | -956.0 (4190.6) | 1180.0 (311.1) | -8281.3 (13425.6) | 6328.3 (17461.8)
  Week 8 (n=4, 6, 2, 5, 3) | -2322.5 (4827.1) | 836.7 (4104.5) | -5695.0 (8605.5) | -3070.0 (4798.4) | 5195.0 (9724.4)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 Eye Drops Vehicle Group in Japan | CP-690,550 Eye Drops 0.001% Group in Japan | CP-690,550 Eye Drops 0.003% Group in Japan | CP-690,550 Eye Drops 0.005% Group in Japan | Sodium Hyaluronate Eye Drops 0.1% Group in Japan | CP-690,550 Eye Drops Vehicle Group in Korea | CP-690,550 Eye Drops 0.001% Group in Korea | CP-690,550 Eye Drops 0.003% Group in Korea | CP-690,550 Eye Drops 0.005% Group in Korea
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42 | 2/41 | 0/40 | 0/39 | 0/21 | 0/19 | 1/21 | 0/21
Other Adverse Events (participants affected / at risk) | 11/41 | 11/42 | 16/41 | 8/40 | 9/39 | 6/21 | 7/19 | 6/21 | 8/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 Eye Drops Vehicle Group in Japan (N=41) | CP-690,550 Eye Drops 0.001% Group in Japan (N=42) | CP-690,550 Eye Drops 0.003% Group in Japan (N=41) | CP-690,550 Eye Drops 0.005% Group in Japan (N=40) | Sodium Hyaluronate Eye Drops 0.1% Group in Japan (N=39) | CP-690,550 Eye Drops Vehicle Group in Korea (N=21) | CP-690,550 Eye Drops 0.001% Group in Korea (N=19) | CP-690,550 Eye Drops 0.003% Group in Korea (N=21) | CP-690,550 Eye Drops 0.005% Group in Korea (N=21)
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 Eye Drops Vehicle Group in Japan (N=41) | CP-690,550 Eye Drops 0.001% Group in Japan (N=42) | CP-690,550 Eye Drops 0.003% Group in Japan (N=41) | CP-690,550 Eye Drops 0.005% Group in Japan (N=40) | Sodium Hyaluronate Eye Drops 0.1% Group in Japan (N=39) | CP-690,550 Eye Drops Vehicle Group in Korea (N=21) | CP-690,550 Eye Drops 0.001% Group in Korea (N=19) | CP-690,550 Eye Drops 0.003% Group in Korea (N=21) | CP-690,550 Eye Drops 0.005% Group in Korea (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival erosion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 2
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Keratitis (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Keratopathy (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meibomian gland dysfunction (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Salivary gland pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenoviral conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 4 | 2 | 5 | 1 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
High density lipoprotein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Optic nerve cup/disc ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.